CLINICAL TRIAL: NCT01676103
Title: The Effects of Supplementing Tyrosine on Blood Pressure in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHS-797
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease (PD); Orthostatic hypotension (OH)
MeSH Terms: conditions — Parkinson Disease; Hypotension, Orthostatic | interventions — Tyrosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tyrosine (Experimental): Tyrosine supplementation (500 mg 2x daily) for 7 days
  Interventions: Dietary Supplement: Tyrosine
- Sugar pill (Placebo Comparator): Placebo sugar pills (2x daily) for 7 days
  Interventions: Other: Placebo Comparator:Sugar Pill

INTERVENTIONS:
Dietary Supplement: Tyrosine — Tyrosine supplementation (500 mg 2 x daily) for 7 days
  Arms: Tyrosine
Other: Placebo Comparator:Sugar Pill — Placebo sugar pills (2x daily
  Arms: Sugar pill

SUMMARY:
The objective of this experiment is:

* Primary: To determine the effects of tyrosine supplementation on orthostatic hypotension in people with PD.
* Secondary: To determine the effects of tyrosine supplementation in people with PD with autonomic insufficiency on HR, BP, and norepinephrine responses during acute exercise stress.

Orthostatic hypotension and autonomic abnormalities are a common problem for individuals who suffer from PD, especially as it leads to lightheadedness and falling. For those affected, it can drastically reduce quality of life. It has been hypothesized that tyrosine may impact upon individuals suffering from PD. There is ample evidence in animal models that supports our theory; however there is no clinical evidence of the impact tyrosine supplementation may have in PD patients who suffer from orthostatic hypotension and blunted BP and HR responses. Positive findings that supplemental tyrosine increases BP and HR in people with PD during daily activities such as standing up from a chair and walking can lead to new therapies to improve Parkinsonian orthostatic hypotension.

Hypothesis We will test the hypothesis that symptomatic individuals with PD on dopamine therapy who suffer from orthostatic hypotension and blunted HR and BP responses will improve after tyrosine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the UK Brain Bank Diagnostic criteria
* Diagnosis of orthostatic hypotension according to EFNS guidelines
* Able to walk on a treadmill comfortably for 6-10 minutes
* Currently taking levodopa
* Subjects between the age of 50-80 years old

Exclusion Criteria:

* Currently taking an amino acid supplement
* Currently taking medication that affects BP
* Normal BP response to testing

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Determine the effects of tyrosine supplementation on orthostatic hypotension in people with PD | 7 days
  Orthostatic Blood Pressure Testing:
  Subjects will sit and rest for 10 minutes. Blood pressure will be taken in this resting position after the 10 minutes. Subjects will then stand upright for 3 minutes. Blood pressure will be taken every minute for those 3 minutes. A drop in systolic BP of 20 mmHg and a 10 mmHg in diastolic drop within these 3 minutes indicates orthostatic hypotension according to the American Academy of Neurology.
  Blood Samples:
  Norepinephrine and tyrosine will all be examined via blood samples drawn by a medical assistant or physician from the forearm vein in vacutainer tubes. Two vacutainers of three cc's of blood will be collected and frozen until analyzed.

SECONDARY OUTCOMES:
To determine the effects of tyrosine supplementation in people with PD with autonomic insufficiency on heart rate, blood pressure, and norepinephrine responses during acute exercise stress. | 7 days
  An exercise stress test using a Modified Bruce Protocol, which consists of five 3-minute stages on a treadmill, will be used to implement acute stress. During the test, heart rate, oxygen consumption (VO2), Respiratory Exchange Ratio (RER), and 12 lead EKG tracings will be recorded at 1-minute intervals and BP and a rate of perceived exertion (RPE) will be recorded. The treadmill test will conclude when subjects attain peak exercise. Peak exercise will be determined when a subject attains any one of the following: 1) 85% of target heart rate; 2) an RPE of 8; 3) inability to maintain the pace of the treadmill; 4) an RER of over 1.3. Additionally, the American College of Sports Medicine (ACSM) guidelines for terminating exercise testing will be followed.
  Subjects will be tested on the first visit and then receive supplementation or placebo for 2x daily for 7 days. Subjects will then repeat all the tests they performed on the first visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne DiFrancisco-Donoghue, PhD, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institue of Technology, Old Westbury, New York, United States

REFERENCES:
- [Background] Barbic F, Perego F, Canesi M, Gianni M, Biagiotti S, Costantino G, Pezzoli G, Porta A, Malliani A, Furlan R. Early abnormalities of vascular and cardiac autonomic control in Parkinson's disease without orthostatic hypotension. Hypertension. 2007 Jan;49(1):120-6. doi: 10.1161/01.HYP.0000250939.71343.7c. Epub 2006 Nov 13. PMID 17101845
- [Background] Kujawa K, Leurgans S, Raman R, Blasucci L, Goetz CG. Acute orthostatic hypotension when starting dopamine agonists in Parkinson's disease. Arch Neurol. 2000 Oct;57(10):1461-3. doi: 10.1001/archneur.57.10.1461. PMID 11030798
- [Background] Goldstein DS, Holmes CS, Dendi R, Bruce SR, Li ST. Orthostatic hypotension from sympathetic denervation in Parkinson's disease. Neurology. 2002 Apr 23;58(8):1247-55. doi: 10.1212/wnl.58.8.1247. PMID 11971094
- [Background] Sharabi Y, Goldstein DS. Mechanisms of orthostatic hypotension and supine hypertension in Parkinson disease. J Neurol Sci. 2011 Nov 15;310(1-2):123-8. doi: 10.1016/j.jns.2011.06.047. Epub 2011 Jul 16. PMID 21762927
- [Background] Karobath M, Diaz JL, Huttunen MO. The effect of L-dopa on the concentrations of tryptophan, tyrosine and serotonin in rat brain. Eur J Pharmacol. 1971 May;14(4):393-6. doi: 10.1016/0014-2999(71)90195-6. No abstract available. PMID 5157767
- [Background] Growdon JH, Melamed E, Logue M, Hefti F, Wurtman RJ. Effects of oral L-tyrosine administration on CSF tyrosine and homovanillic acid levels in patients with Parkinson's disease. Life Sci. 1982 Mar 8;30(10):827-32. doi: 10.1016/0024-3205(82)90596-3. PMID 6175872
- [Background] Glaeser BS, Melamed E, Growdon JH, Wurtman RJ. Elevation of plasma tyrosine after a single oral dose of L-tyrosine. Life Sci. 1979 Jul 16;25(3):265-71. doi: 10.1016/0024-3205(79)90294-7. No abstract available. PMID 481129
- [Background] Stryjer R, Klein C, Treves TA, Rabey JM. The effects of acute loading with levodopa and levodopa with selegiline on blood pressure and plasma norepinephrine levels in chronic Parkinson's disease patients. Acta Neurol Scand. 2005 Feb;111(2):89-94. doi: 10.1111/j.1600-0404.2005.00294.x. PMID 15644067
- [Background] Tipre DN, Goldstein DS. Cardiac and extracardiac sympathetic denervation in Parkinson's disease with orthostatic hypotension and in pure autonomic failure. J Nucl Med. 2005 Nov;46(11):1775-81. PMID 16269589
- [Background] Riederer P. L-dopa competes with tyrosine and tryptophan for human brain uptake. Nutr Metab. 1980;24(6):417-23. doi: 10.1159/000176359. PMID 7219901
- [Background] Deijen JB, Orlebeke JF. Effect of tyrosine on cognitive function and blood pressure under stress. Brain Res Bull. 1994;33(3):319-23. doi: 10.1016/0361-9230(94)90200-3. PMID 8293316
- [Background] Conlay LA, Maher TJ, Wurtman RJ. Tyrosine increases blood pressure in hypotensive rats. Science. 1981 May 1;212(4494):559-60. doi: 10.1126/science.7209553.
- [Background] Conlay LA, Maher TJ, Wurtman RJ. Tyrosine accelerates catecholamine synthesis in hemorrhaged hypotensive rats. Brain Res. 1985 Apr 29;333(1):81-4. doi: 10.1016/0006-8993(85)90126-x. PMID 3995291
- [Background] Lahrmann H, Cortelli P, Hilz M, Mathias CJ, Struhal W, Tassinari M. EFNS guidelines on the diagnosis and management of orthostatic hypotension. Eur J Neurol. 2006 Sep;13(9):930-6. doi: 10.1111/j.1468-1331.2006.01512.x. PMID 16930356
- [Background] DiFrancisco-Donoghue J, Elokda A, Lamberg EM, Bono N, Werner WG. Norepinephrine and cardiovascular responses to maximal exercise in Parkinson's disease on and off medication. Mov Disord. 2009 Sep 15;24(12):1773-8. doi: 10.1002/mds.22612. PMID 19562762
- [Derived] DiFrancisco-Donoghue J, Rabin E, Lamberg EM, Werner WG. Effects of Tyrosine on Parkinson's Disease: A Randomized, Double-Blind, Placebo-Controlled Trial. Mov Disord Clin Pract. 2014 Oct 23;1(4):348-353. doi: 10.1002/mdc3.12082. eCollection 2014 Dec. PMID 30363894